CLINICAL TRIAL: NCT04981990
Title: Single Lung Ventilation Versus Two Lung Ventilation in Video Assisted Lung Surgeries
Brief Title: Single Lung Ventilation Versus Two Lung Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Esraa Abdellatif, Anesthesia resident, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Anesth
Record Dates: First submitted 2021-04-22; First posted 2021-07-29 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Hypoxemia; Single Lung Ventilation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Two equal groups: the first group undergoing lung surgeries with single lung ventilation by double lumen endotracheal tube, the second group undergoing lung surgeries with two lung ventilation using conventional single lumen endotracheal tube
Who Masked: Participant
Masking Description: The patients will not know whether they are in the first or second group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single lung ventilation (Active Comparator): Using double lumen endotracheal tube and lung isolation
  Interventions: Procedure: Single lung ventilation by double lumen endotracheal tube
- Two lung ventilation (Active Comparator): Using conventional single lumen endotracheal tube and intermittent two lung ventilation
  Interventions: Procedure: Two lung ventilation by conventional single lumen endotracheal tube

INTERVENTIONS:
Procedure: Single lung ventilation by double lumen endotracheal tube — Single lung ventilation using double lumen endotracheal tube and isolation of the operated lung during surgery to create ideal surgical field
  Arms: Single lung ventilation
Procedure: Two lung ventilation by conventional single lumen endotracheal tube — Intermittent two lung ventilation so that no significant hypoxia occurs with creating optimum surgical field
  Arms: Two lung ventilation

SUMMARY:
Hypoxia in single lung ventilation versus two lung ventilation in video assisted lung surgeries

DETAILED DESCRIPTION:
Incidence of hypoxia in single lung ventilation by double lumen endotracheal tube "of choice in lung surgeries" versus incidence of hypoxia in two lung ventilation by conventional single lumen endotracheal tube "intermittent two lung ventilation"

ELIGIBILITY:
Inclusion Criteria:

* Age group: Adult patients from age of 21 years to 60 years
* Sex: Both sexes
* ASA Classification: patients with ASA classification II, III.
* Elective lung surgeries using video assisted thoracoscopic surgeries.

Exclusion Criteria:

* Patients refuse to give informed consent.
* ASA Classification: ASA IV.
* Failure of thoracoscopic surgeries and continue as open thoracotomy
* Patients with ischemic heart diseases, where hypoxemia might be preexisting, or patient be more vulnerable to hypoxemia whatever the technique or time of hypoxia.
* Emergency lung surgeries.
* Patients underwent previous lung surgeries of any cause.
* Patients with pathology to the non-operated side.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxemia | Intraoperative to first 24 hours post operative
  Hypoxemia in single and two lung ventilation by serial arterial blood gases

SECONDARY OUTCOMES:
Incidence of failure to correct Hypoxemia in single lung ventilation | Intraoperative
  Stop lung isolation and procedure using two lung ventilation to correct hypoxia
Incidence of failure of two lung ventilation to create optimum surgical field | Intraoperative
  Frequent stopping of ventilation and the surgent can't access the surgical field easily
Incidence of post operative complications | First 24 hours post operative
  Any associated complications

CONTACTS AND LOCATIONS:
Overall Officials: Esraa Abdellatif, M.B., B.Ch., Principal Investigator — Anesthesiology department; Omar El safty, MD, Study Chair — Anesthesiology department; Salwa Omar, MD, Study Director — Anesthesiology department; Mohamed Taeimah, MD, Study Director — Anesthesiology department
Locations (1):
- Aun Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All study data will be open to other researchers
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After finishing the study by the end of August 2021
Access Criteria: For any medical student or staff interested in topic without any other considerations

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT04981990/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT04981990/ICF_001.pdf